CLINICAL TRIAL: NCT05698797
Title: Effects of Proprioceptive Training vs. Hip Abductor With External Rotator Strengthening on Pain and Functions in Patients With Patellofemoral Pain Syndrome
Brief Title: Proprioceptive Training vs. Hip Abductor With External Rotator Strengthening in Patients With Patellofemoral Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AWH/EC/03/2021
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Hip muscles strengthening; Rehabilitation; Proprioceptive training; Exercises
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (Experimental): In this group participants received hip abductor and external rotator strengthening exercises in addition to conventional physical therapy.
  Interventions: Other: Hip strengthening exercises
- Experimental group 2 (Active Comparator): In this group participants received proprioceptive training and conventional physical therapy.
  Interventions: Other: Proprioceptive training
- Control group (Active Comparator): In this group participants received conventional physical therapy alone.
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Hip strengthening exercises — Hip abductor and external rotator strengthening exercises were performed for 4 weeks.
  Arms: Experimental group 1
Other: Proprioceptive training — Proprioceptive training consisted of eight exercises was performed for 4 weeks.
  Arms: Experimental group 2
Other: Conventional physical therapy — Conventional physical therapy included interferential therapy and two types of knee-strengthening exercises.
  Arms: Control group

SUMMARY:
Patellofemoral pain syndrome (PFPS) is a common musculoskeletal disorder characterized by an insidious onset of pain in the knee's anterior /retro-patellar / peripatellar region. Even though various rehabilitation approaches, including hip strengthening and proprioceptive training, are being considered for managing PFPS, the most appropriate treatment from these two is still unclear. Therefore, this study aimed to compare the program consisting of hip abductors and external rotators strengthening exercises vs. the program consisting of proprioceptive training of the knee to identify the most effective rehabilitation approach for patients suffering from PFPS.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years
* Patients diagnosed recently by an orthopedic surgeon for Patello-femoral pain syndrome
* experiencing anterior/retro patellar knee pain during activities,
* insidious onset of symptoms not linked to trauma,
* pain persisting for no less than four weeks,
* pain on palpation of the patellar facets,
* pain when stepping down from a 25-cm step or during a double-legged squat.

Exclusion Criteria:

* Patients with recent lower limb fractures or dislocations,
* knee/hip joint surgery,
* signs, symptoms, or radiological findings of intra-articular pathology such as effusion, ligamentous or meniscal involvement,
* those with indications of patellar apprehension,
* referred pain from the hip, back, or sacroiliac joint,
* acute knee strain or sprain,
* on medication such as NSAIDs or corticosteroids,
* degenerative and infectious arthritis

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Kujala Anterior Knee Pain Scale (AKPS) | 4 weeks.
  Pain was measured using the AKPS. The AKPS is scored from a minimum score of 0 to a maximum score of 100 points. Lower scores indicate greater pain and disability.

CONTACTS AND LOCATIONS:
Overall Officials: Masood Khan, M.P.Th, Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raju A, Jayaraman K, Nuhmani S, Sebastian S, Khan M, Alghadir AH. Effects of hip abductor with external rotator strengthening versus proprioceptive training on pain and functions in patients with patellofemoral pain syndrome: A randomized controlled trial. Medicine (Baltimore). 2024 Feb 16;103(7):e37102. doi: 10.1097/MD.0000000000037102. PMID 38363950